CLINICAL TRIAL: NCT00117910
Title: An Open Label, Randomised, Multicentre Study of Pegfilgrastim in Primary Versus Secondary Prophylaxis of Neutropenia as an Adjunct to Chemotherapy in Elderly Subjects With High Risk Breast Cancer.
Brief Title: Treatment for Elderly Patients With High Risk Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20020106
Record Dates: First submitted 2005-06-30; First posted 2005-07-11 (Estimated); Last update posted 2008-05-16 (Estimated); Status verified 2008-05

CONDITIONS: Breast Cancer
Keywords: Aged, Granulocyte Colony-Stimulating Factor; Combined Modality Therapy, Neutropenia; pegfilgrastim, Neulasta®; FEC-100, Antineoplastic Agents; Breast Cancer, Female
MeSH Terms: conditions — Breast Neoplasms; Neutropenia | interventions — pegfilgrastim

INTERVENTIONS:
Drug: pegfilgrastim

SUMMARY:
This open-label, multicenter study explored primary and secondary prophylaxis treatment with a single, fixed-dose, subcutaneous (SC) injection of pegfilgrastim in elderly subjects with high-risk breast cancer receiving myelosuppressive chemotherapy. The primary objective was to provide preliminary information on the incidence of protocol defined neutropenic events in chemotherapy cycle 1.

ELIGIBILITY:
Inclusion Criteria: - High-risk, stage II-III breast cancer suitable for treatment with up to 6 cycles of FEC-100 - Chemotherapy - Histologically proven greater than or equal to 1 axillary nodes positive - Oestrogen receptor negative or positive - Chemotherapy naïve - VES 13 (Vulnerable Elders Survey) score less than or equal to 3 - ECOG performance status less than or equal to 2 - ANC greater than or equal to 1.5 x 10^9/L - Platelets greater than or equal to 100 x 10^9/L - Adequate renal function (serum creatinine less than 1.5 x upper limit of normal (ULN)) - Before any study specific procedure the subject must give written informed consent for participation in the study Exclusion Criteria: - Total serum bilirubin greater than ULN according to institutional standard - Clinically significant cardiac disease that would preclude the use of epirubicin (e.g., LVEF (left ventricular ejection fraction)) less than 45% at rest by MUGA or echocardiogram - Prior bone marrow or stem cell transplantation - Any premalignant myeloid condition or any malignancy with myeloid characteristics (e.g., myelodysplastic syndromes, acute or chronic myelogenous leukaemia) - History of prior malignancy other than breast cancer with the exception of curatively treated basal cell carcinoma, in situ cervical carcinoma or surgically cured malignancies - Prior radiation therapy - Active infection or administration of systemic antibiotics or anti-infectives within 72 hours before start of chemotherapy - Known hypersensitivity to E coli-derived products (e.g., Filgrastim, HUMULIN®, Insulin, L-Asparaginase, HUMATROPE®, Growth Hormone, INTRON A®) - Previous exposure to pegfilgrastim or previous entry into this study - Known HIV infection - Inability to understand the nature of the study and provide written informed consent - Subject currently enrolled in another investigational device or drug trial(s) or has received other investigational agent(s), with the exception of placebo-treated subjects, within the last 30 days - Concerns for subject's compliance with the protocol procedures

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Dates: Start 2002-10; Study Completion 2004-05

PRIMARY OUTCOMES:
Provide preliminary information on the incidence of protocol defined neutropenic events in chemotherapy cycle 1.

SECONDARY OUTCOMES:
Provide preliminary information on primary and secondary prophylaxis treatment with pegfilgrastim with respect to:
Incidence of protocol defined neutropenic events over all cycles
Incidence of dose reductions and dose delays of planned chemotherapy due to
hematological toxicity
Relative dose intensity
Safety profile over all cycles

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Romieu G, Clemens M, Mahlberg R, Fargeot P, Constenla M, Schutte M, Easton V, Skacel T, Bacon P, Brugger W. Pegfilgrastim supports delivery of FEC-100 chemotherapy in elderly patients with high risk breast cancer: a randomized phase 2 trial. Crit Rev Oncol Hematol. 2007 Oct;64(1):64-72. doi: 10.1016/j.critrevonc.2006.12.007. Epub 2007 Feb 20. PMID 17317205
- [Derived] Brugger W, Bacon P, Lawrinson S, Romieu G. Neutrophil recovery in elderly breast cancer patients receiving adjuvant anthracycline-containing chemotherapy with pegfilgrastim support. Crit Rev Oncol Hematol. 2009 Dec;72(3):265-9. doi: 10.1016/j.critrevonc.2009.05.002. Epub 2009 Oct 23. PMID 19596586
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_11_GCSFSD01_20020106.pdf
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com